CLINICAL TRIAL: NCT03358199
Title: Laparoscopic Ovarian Drilling Before IVF/ICSI in Polycystic Ovarian Syndrome Patients With High Antimullarian Hormone
Brief Title: LOD Before IVF/ICSI in PCOS Patients With High AMH
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Abdelhafez, Principal Investigator, Mansoura University
Other Study IDs: MSA6
Record Dates: First submitted 2017-11-27; First posted 2017-11-30 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Infertility; Polycystic Ovarian Syndrome
Keywords: LOD; PCOS; AMH; OHSS
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: PCOS women with AMH level (≥ 7 ng/ml) who underwent LOD in the preceding 3 months prior to IVF/ICSI
  Interventions: Procedure: LOD
- Control group: PCOS women with AMH level (≥ 7 ng/ml) who did not undergo LOD in the preceding 3 months prior to IVF/ICSI

INTERVENTIONS:
Procedure: LOD — Women underwent LOD in the preceding 3 months prior to IVF/ICSI
  Other Names: Laparoscopic ovarian drilling
  Groups: Study group

SUMMARY:
To evaluate the effect of performing laparoscopic ovarian drilling (LOD) before proceeding to in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) on the cycle outcomes in polycystic ovarian syndrome (PCOS) patients with high antimullerian hormone (AMH) levels

DETAILED DESCRIPTION:
Retrospective case-control study of PCOS women with high serum AMH level (≥ 7 ng/ml) who were subjected IVF/ICSI. Women underwent LOD in the preceding 3 months prior to IVF/ICSI (study group) will be compared with a control group of women who did not underwent LOD (control group)

ELIGIBILITY:
Inclusion Criteria:

* PCOS women subjected to COS through fixed gonadotropin releasing hormone (GnRH) antagonist protocol with final triggering of oocyte maturation by GnRH agonist (GnRHa)
* Elevated serum AMH level (≥ 7 ng/ml)

Exclusion Criteria:

* Age < 18 years or > 35 years
* Body mass index (BMI) < 19 kg/m2 or > 35 kg/m2
* Use of cabergoline therapy or coasting to minimize the risk of OHSS

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fertility care clinic
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-03-22 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-18 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 36-38 hours after triggering of oocyte maturation
  Number of collected oocytes during oocyte retrieval
Oocyte maturity rate | Within one hour after oocyte retrieval
  Calculated for each woman by dividing the number of mature oocytes (MII oocytes) by the total number of oocytes retrieved
Fertilization rate | 20-24 hours after injection (or insemination)
  Calculated for each couple by dividing the number of fertilized oocytes by the number of injected (or inseminated) oocytes

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6 weeks after embryo transfer
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 4-6 weeks after the ET) divided by the number of ET procedures
Implantation rate | 6 weeks after embryo transfer
  Number of gestational sacs on TVS scan at 4-6 weeks after ET divided by the number of transferred embryos
Incidence of early OHSS | Within 9 days of final triggering of oocyte maturation
  Incidence of OHSS within 9 days of final triggering of oocyte maturation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Abdelhafez, Dr, Principal Investigator — Mansoura University; Alaa Wageh, Dr, Study Director — Mansoura University; Waleed El-refaie, Dr, Study Director — Mansoura University; Maher Shams, Dr, Study Director — Mansoura University
Locations (1):
- Fertility Care Unit (FCU) in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided